CLINICAL TRIAL: NCT07226986
Title: A Phase Ib/II Open-label, Multi-center Study of AMO959 With Lutetium (177Lu) Vipivotide Tetraxetan (AAA617) in Combination With an Androgen Receptor Pathway Inhibitor (ARPI) in Adult Participants With PSMA-positive Metastatic Castration Resistant Prostate Cancer (mCRPC)
Brief Title: A Phase Ib/II Open-label Study of AMO959 With Lutetium (177Lu) Vipivotide Tetraxetan (AAA617) in Combination With ARPI in Adult Participants With PSMA-positive mCRPC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAMO959A12103; 2025-521859-23-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2025-11-07; First posted 2025-11-12 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: PSMA-positive Metastatic Castration Resistant Prostate Cancer (mCRPC) With Prior Exposure to One Prior ARPI Who Are Candidates for Taxane-based Chemotherapy
Keywords: PSMA-positive metastatic castration resistant prostate cancer; AMO959; Lutetium (177Lu) vipivotide tetraxetan; Androgen Receptor Pathway Inhibitor (ARPI); dose escalation
MeSH Terms: interventions — Pluvicto; enzalutamide; abiraterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 1b: Doublet (Experimental): Participants will receive AMO959 BID for first 14 days followed by AAA617+AMO959 every 6 weeks for a maximum of 6 cycles.
  Interventions: Drug: AMO959; Radiation: AAA617
- Phase 1b: Triplet (Experimental): Participants will receive AAA617 on day 1 followed by AMO959 BID (days 2-15), repeated every 6 weeks, for a maximum of 6 cycles with an ARPI (abiraterone or enzalutamide) administered continuously starting on day 1.
  Interventions: Drug: AMO959; Radiation: AAA617; Drug: Enzalutamide; Drug: Abiraterone
- Phase 1b: Food Effect (Experimental): Participants will receive a single dose of AMO959 on Day 1 (fed), followed by 2-day washout, then AMO959 BID (fasted) for 14 days followed by 2-day washout and AAA617+AMO959 (fasted) every 6 weeks for a maximum of 6 cycles.
  Interventions: Drug: AMO959; Radiation: AAA617
- Phase II: Arm 1 (Experimental): Participants will receive AAA617 on day 1 followed by AMO959 BID (days 2-15), repeated every 6 weeks, for a maximum of 6 cycles with an ARPI (abiraterone or enzalutamide administered continuously starting on day 1.
  Interventions: Drug: AMO959; Radiation: AAA617; Drug: Enzalutamide; Drug: Abiraterone
- Phase II: Arm 2 (Experimental): Participants will receive AAA617 on day 1 followed by AMO959 BID (days 2-15), repeated every 6 weeks, for a maximum of 6 cycles with an ARPI (abiraterone or enzalutamide) administered continuously starting on day 1.
  Interventions: Drug: AMO959; Radiation: AAA617; Drug: Enzalutamide; Drug: Abiraterone
- Phase II: Arm 3 (Experimental): Participants will receive AAA617 every 6 weeks for a maximum of 6 cycles, with ARPI (abiraterone or enzalutamide) administered continuously starting on day 1.
  Interventions: Radiation: AAA617; Drug: Enzalutamide; Drug: Abiraterone

INTERVENTIONS:
Drug: AMO959 — DNA Damage Response inhibitor
  Other Names: BY1298; BY101298
  Arms: Phase 1b: Doublet; Phase 1b: Food Effect; Phase 1b: Triplet; Phase II: Arm 1; Phase II: Arm 2
Radiation: AAA617 — PSMA-targeted radiopharmaceutical
  Other Names: Pluvicto [177Lu]Lu-PSMA-617
Drug: Enzalutamide — Androgen receptor pathway inhibitor
  Arms: Phase 1b: Triplet; Phase II: Arm 1; Phase II: Arm 2; Phase II: Arm 3
Drug: Abiraterone — Androgen receptor pathway inhibitor
  Arms: Phase 1b: Triplet; Phase II: Arm 1; Phase II: Arm 2; Phase II: Arm 3

SUMMARY:
The purpose of this phase Ib/II study is to (a) in Phase Ib evaluate the safety, tolerability, and pharmacokinetics (PK) of AMO959 when given in combination with lutetium (177Lu) vipivotide tetraxetan (also known as [177Lu]Lu-PSMA-617 or 177Lu-PSMA-617 and hereafter referred to as AAA617) with an androgen receptor pathway inhibitor (ARPI) in participants with metastatic castration resistant prostate cancer (mCRPC) who have failed one prior ARPI and with or without prior taxane exposure, and (b) in Phase II evaluate the preliminary efficacy of AMO959 in combination with AAA617 and ARPI in participants with mCRPC who have failed one prior ARPI, but who have not yet been exposed to taxane treatment.

DETAILED DESCRIPTION:
This study will consist of two phases:

1. The escalation phase (Ib) will consist of provisionally three dose level cohorts of 3-6 participants investigating the safety, tolerability, and to determine the recommended dose for expansion (RDE) of AMO959 with standard dose of AAA617 +/- ARPI (abiraterone or enzalutamide). Initially AMO959 monotherapy will be administered, and then AMO959 will be given along with AAA617 in the same participants. Dose escalation meetings (DEMs) will occur when all participants in a dose level cohort have completed the DLT evaluation period or have experienced a DLT prior to the end of the evaluation period.
2. The Phase II will follow with 25 participants per arm randomized in a 1:1:1 ratio treated at the RDE(s) of AMO959 along with AAA617 and ARPI (abiraterone or enzalutamide) and AAA617 and ARPI (abiraterone or enzalutamide).

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Participants must be adults ≥ 18 years of age.
* Participants must have an ECOG performance status of 0 to 2.
* Participants must have histologically confirmed adenocarcinoma of the prostate. Participants with other histology (e.g. neuroendocrine, intraductal subtype) are not eligible.
* Phase Ib: Prior exposure of up to 1 line of taxane-based chemotherapy is permissible. Phase II: Participants must not have received taxane-based chemotherapy in mCRPC setting (allowed in mHSPC setting).
* Participants must have PSMA-PET positive disease assessed by using a PSMA imaging agent that is approved as per protocol and are eligible as determined by the sponsor's central reading rules.
* Castration level of testosterone (< 50 ng/dL), and/or use of concomitant ADT
* Participant must have been diagnosed with mCRPC with documented progressive disease while on treatment with ARPI in mHSPC or earlier setting as their last treatment (and did not progress on more than one ARPI), based on at least 1 of the following criteria:

  * Serum/plasma PSA progression is defined as 2 increases in PSA measured at least 1 week apart. The minimal start value is 2.0 ng/mL; 1.0 ng/mL is the minimal starting value if confirmed rise in PSA is the only indication of progression as per PCWG3 guidelines.
  * Soft-tissue progression defined PCWG3-modified RECIST v1.1 (Eisenhauer et al 2009, Scher et al 2016).
  * Progression of bone disease: 2 new lesions; only positivity on the bone scan defines metastatic disease to bone (PCWG3 criteria Scher et al 2016).

Key Exclusion Criteria:

* Concurrent local (radiation therapy to the prostate with curative intent or other prostate antineoplastic ablative procedures) or systemic (hormonal ablation, chemotherapy, immunotherapy, , RLTs) antineoplastic treatments, or within 28 days of enrollment (Phase Ib) or randomization (Phase II)
* Prior treatment with any RLT or PSMA-targeted agents (approved or investigational)
* Any other investigational agents within 28 days prior to first dose of any study treatment
* Concurrent serious medical conditions that may interfere with study procedures or followup
* Participants with a history of CNS metastases must have received therapy (surgery, whole brain radiation therapy, stereotactic radiosurgery) and be neurologically stable, asymptomatic, and not taking corticosteroids for the purpose of maintaining neurologic integrity.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2028-07-10 (Estimated); Study Completion 2029-09-13 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Incidence rate of Dose-limiting toxicities (DLTs) | Up to 42 days after the first AAA617 dose administration
  Incidence of dose limiting toxicities (DLTs) with AMO959 in combination with AAA617 +/- ARPI A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness/injury, or concomitant medications that occurs within the evaluation period and meets any of the criteria specified in the protocol. The National Cancer Institute Common Terminology Criteria for Adverse events (NCI CTCAE) version 5.0 will be used for all grading.
Phase Ib: Incidence rate of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From date of start of study treatment, assessed up to approximately 45 months
  Incidence of adverse events by type, frequency, and severity, as graded by the NCI CTCAE version 5.0.
Phase Ib: Number of Participants with dose adjustments | From date of start of study treatment, assessed up to approximately 24 months
  The number of participants with dose adjustments (reductions, interruption, or permanent discontinuation).
Phase Ib: Dose Intensity | From date of start of study treatment, assessed up to approximately 24 months
  Dose intensity (computed as the ratio of actual cumulative dose received and actual duration of exposure) and the relative dose intensity (computed as the ratio of dose intensity and planned dose intensity).
Phase Ib: Duration of exposure to each study drug | From date of start of study treatment, assessed up to approximately 24 months
  Duration of exposure (in months) to each study drug.
Phase II: Biochemical Response (PSA50) | From date of start of study treatment, assessed up to approximately 24 months
  Biochemical response (PSA50), defined as the proportion of participants who achieved a ≥ 50% decrease in PSA from baseline at any time during the treatment period prior to start of new anti-cancer therapy that is confirmed by a second PSA measurement ≥ 4 weeks later.

SECONDARY OUTCOMES:
Prostate Specific Antigen 90 (PSA90) response | From date of start of study treatment, assessed up to approximately 24 months
  PSA90 response is defined as the proportion of participants who have achieved a ≥ 90% decrease in PSA from baseline at any time during the treatment period prior to start of new anti-cancer therapy that is confirmed by a second PSA measurement ≥4 weeks later.
Phase Ib: Prostate Specific Antigen 50 (PSA50) response | From date of start of study treatment, assessed up to approximately 24 months
  PSA50 response is defined as the proportion of participants who have achieved a ≥ 50% decrease in PSA from baseline at any time during the treatment period prior to the start of new anti-cancer therapy, confirmed by a second PSA measurement ≥4 weeks later.
Phase Ib and Phase II: Radiographic progression-free survival (rPFS) | From date of start of study treatment (Phase Ib) / randomization (Phase II), assessed up to approximately 24 months
  Radiographic progression- free survival (rPFS) is defined as the time from the date of start of study treatment (Phase Ib) / randomization (Phase II) to the date of first documented radiographic disease progression using conventional imaging and Prostate Cancer Working Group 3 (PCWG3)-modified RECIST v1.1 criteria (Scher et al 2016) or death due to any cause, whichever occurs first.
Phase Ib and Phase II: Overall Response Rate (ORR) | From date of start of study treatment (Phase Ib) / randomization (Phase II), assessed up to approximately 24 months
  Overall Response Rate (ORR) is defined as the proportion of participants with best overall response (BOR) of confirmed complete response (CR) or partial response (PR) in soft tissue based on tumor response data and according to PCWG3-modified RECIST v1.1, in the absence of bone progression as per PCWG3.
Phase Ib and Phase II: Disease control rate (DCR) | From date of start of study treatment (Phase Ib) / randomization (Phase II), assessed up to approximately 24 months
  Disease control rate (DCR) is defined as the proportion of participants with a BOR of confirmed CR or PR, stable disease (SD) or Non-CR/Non- progressive disease (PD) in soft tissue based on tumor response data and according to PCWG3-modified RECIST v1.1, in the absence of bone progression as per PCWG3.
Phase Ib and Phase II: Duration of Response (DoR) | From date of start of study treatment (Phase Ib) / randomization (Phase II), assessed up to approximately 24 months
  Duration of Response (DoR) is defined as the duration of time between the date of first documented response (CR or PR) according to PCWG3- modified RECIST v1.1, in the absence of bone progression as per PCWG3, based on tumor response data and the date of first documented radiographic progression in soft tissue or death due to any cause, whichever occurs first.
Overall Survival (OS) | From date of start of study, assessed up to approximately 45 months
  Overall Survival (OS) is defined as the time from the date of start of study treatment (Phase Ib) / randomization (Phase II) to the date of death due to any cause.
Phase II: Time to soft tissue progression (TTSTP) | From date of start of study randomization, assessed up to approximately 24 months
  Time to soft tissue progression (TTSTP) is defined as time from randomization to the date of first documented radiographic soft tissue progression per PCWG3-modified RECIST v1.1.
Phase Ib: Plasma concentrations of AMO959 | Throughout run-in periods and first cycle with AAA617, assessed up to 6 months
  AMO959 pharmacokinetic (PK) samples will be obtained and evaluated in all participants at all dose levels by treatment arms
Phase Ib: Plasma concentrations of AAA617 | Throughout treatment periods with AAA617, assessed up to 6 months
  AAA617 pharmacokinetic (PK) samples will be obtained and evaluated in all participants at all dose levels by treatment arms
Phase Ib: Time activity curves (TACs) for AAA617 | Throughout treatment periods with AAA617, assessed up to 6 months
  Time Activity Curves (TAC) will be generated by plotting concentrations against time.
Phase Ib: Absorbed radiation doses in selected organs and tumor lesions for AAA617 | Throughout treatment periods with AAA617, assessed up to 6 months
  The organ absorbed radiation dose and effective radiation dose will be evaluated.
Phase II: Incidence rate of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From date of start of study treatment, assessed up to approximately 45 months
  Incidence of adverse events by type, frequency, and severity, as graded by the NCI CTCAE version 5.0.
Phase II: Number of Participants with dose adjustments | From date of start of study treatment, assessed up to approximately 24 months
  The number of participants with dose adjustments (reductions, interruption, or permanent discontinuation).
Phase II: Dose Intensity | From date of start of study treatment, assessed up to approximately 24 months
  Dose intensity (computed as the ratio of actual cumulative dose received and actual duration of exposure) and the relative dose intensity (computed as the ratio of dose intensity and planned dose intensity).
Phase II: Duration of exposure to each study drug | From date of start of study treatment, assessed up to approximately 24 months
  Duration of exposure (in months) to each study drug.
Phase II: Radiographic Progression Free Survival (rPFS) by Positron Emission Tomography (PET) (rPFS-PET) | From date of start of study randomization, assessed up to approximately 24 months
  Radiographic Progression Free Survival (rPFS) by Positron Emission Tomography (PET) (rPFS- PET) is defined as the time from the date of randomization to first documented radiographic disease progression (an increase in PSMA-positive tumor volume ≥ 20% from baseline and new PSMA-positive malignant lesions) using PSMA PET/CT imaging (Seifert et al 2023, Gafita et al 2023) or death due to any cause, whichever occurs first.
Phase II: Change from baseline in FACT-P Prostate Cancer Subscale (PCS) | From date of start of study, assessed up to approximately 45 months.
  Change from baseline in FACT-P PCS refers to the difference in a patient's score on the Prostate Cancer Subscale (PCS) of the Functional Assessment of Cancer Therapy-Prostate (FACT-P) questionnaire between the start of a study (baseline) and subsequent time points.
Phase II: Time to worsening on the Brief Pain Inventory - Short Form (BPI-SF) | From date of start of study, assessed up to approximately 45 months.
  Time to worsening on the Worst Pain defined as the time from the date of randomization to the first occurrence of worsening on the Brief Pain Inventory - Short Form (BPI-SF) Worst Pain item of at least 30% increase from baseline or a minimum of 2 points increase from baseline or death due to any cause, whichever occurs first.
Phase II: Time to first symptomatic skeletal event (TTSSE) | From date of start of study randomization, assessed up to approximately 24 months.
  Time to first symptomatic skeletal event (TTSSE) is defined as the time from the date of randomization to the date of first new symptomatic pathological bone fracture, spinal cord compression, tumor-related orthopedic surgical intervention, or requirement for radiation therapy to relieve bone pain, or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Murdoch, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com